CLINICAL TRIAL: NCT03020459
Title: Comparing the Surgical Outcomes of Internal Limiting Membrane Peeling-reposition Versus Peeling in Idiopathic Macular Holes: A Randomized Controlled Trial
Brief Title: Internal Limiting Membrane Peeling-reposition to Treat Idiopathic Macular Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH-16-049
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2019-02

CONDITIONS: Macular Hole; Surgery
Keywords: macular holes
MeSH Terms: conditions — Retinal Perforations | interventions — Tooth Exfoliation; coomassie Brilliant Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peeling-reposition (Experimental): After dying with Brilliant Blue G (Brilliant Blue; Gender, Germany) with the help of Constellation 23-gauge vitrectomy system (Alcon Laboratories Inc, Fort Worth, TX), the intervention of "peeling-reposition" was used to peel and unfold the ILM. And the postoperative posture would be prone position in two weeks for all patients after the operation.
  Interventions: Procedure: peeling-reposition; Drug: Brilliant Blue G; Other: postoperative posture; Device: Constellation 23-gauge vitrectomy system
- peeling (Active Comparator): After dying with Brilliant Blue G (Brilliant Blue; Gender, Germany) with the help of Constellation 23-gauge vitrectomy system, the intervention of "peeling" was used to grasped ILM with end-gripping forceps. And the postoperative posture would be prone position in two weeks for all patients after the operation.
  Interventions: Procedure: peeling; Drug: Brilliant Blue G; Other: postoperative posture; Device: Constellation 23-gauge vitrectomy system

INTERVENTIONS:
Procedure: peeling-reposition — After dying with Brilliant Blue G (BBG, Brilliant Blue; Gender, Germany), a horizontal ILM strip is peeled off in inferior quadrant of macular area. Then the ILM was peeled from inferior to superior area continuously. The" ILM roll " was unfolded with assistance of perfluoro-n-octane (PFO). Finally, the position of the fixed ILM flap is adjusted under PFO bubble using flute needle or forceps.This was followed by a complete fluid-gas exchange using 14% perfluoropropane gas.Patients are introduced to maintain facedown position for two weeks postoperatively.
  Arms: peeling-reposition
Procedure: peeling — After dying with Brilliant Blue G (Brilliant Blue; Gender, Germany), a horizontal ILM strip is peeled off in inferior quadrant of macular area. Then, the strand of ILM was peeled off radially from the foveal center to vascular arcade. In result, a round -shaped with 2.5-3.5 disc diameter ILM -peeled area was created.This was followed by a complete fluid-gas exchange using 14% perfluoropropane gas. Patients are encourage to maintain facedown position for two weeks postoperatively.
  Arms: peeling
Drug: Brilliant Blue G — We intravitreal injected 0.1ml of Brilliant Blue G (Brilliant Blue; Gender, Germany) to dye ILM before ILM peeling.
  Other Names: BBG
Other: postoperative posture — Patients of both two groups need to keep prone position for two weeks after the operation.
Device: Constellation 23-gauge vitrectomy system — All surgical procedures are operated on the Constellation 23-gauge vitrectomy system (Alcon Laboratories Inc, Fort Worth, TX).

SUMMARY:
To compare the morphologic and functional outcomes of internal limiting membrane peeling-reposition versus peeling in idiopathic macular holes

DETAILED DESCRIPTION:
This randomized clinical trial will be performed at a single center. Eligible patients with idiopathic macular holes will be equally randomized to internal limiting membrane (ILM) peeling-reposition group or ILM peeling group through computer-aided random allocation.

A standard 3-port pars plana vitrectomy was performed by a single surgeon using the Constellation 23 gauge vitrectomy system (Alcon Laboratories Inc, Fort Worth, Texas, USA).After posterior vitreous detachment was achieved, peeling of the ILM was performed by an end gripping forceps with the assistance of Brilliant Blue G. In ILM peeling-reposition group, the peeled ILM flap is flatten back to peeled area with assistance of perfluoro-n-octane. In ILM peeling group, a round shape with 2.5 to 3.5 disc diameter of ILM is peeled. This is followed by a complete fluid-gas exchange. Patients are encouraged to maintain a face-down position for two weeks postoperatively in two groups.

Postoperative measurements of BCVA and spectral domain optical coherence tomography(SD-OCT) are conducted at 1,3 and 6-month follow-up visits by independent masked observers. Macular light sensitivity and fixation stability are determined with microperimetry at 1,3, and 6 months of follow-up. Mf-ERG, M-score chart and VFQ-25 chart are performed 1,3, and 6 months of follow-up.

Comparison of BCVA, anatomical closure were primarily performed between the two groups. Then, the morphologic changes of inner retina and the functional parameters measured from microperimetry, Mf-ERG, M-score chart, VFQ-25 chart were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed as macular hole by optical coherence tomography.
* Age ranges from 50 to 80 years.
* The patients have indication for surgery.

Exclusion Criteria:

* Traumatic macular hole.
* Combined with serious epiretinal membrane.
* Combined with diabetic retinopathy, hypertensive retinopathy.
* Combined with other ocular diseases, such as keratitis，uveitis，retinal vasculitis.
* - 6.0 diopters or more of spherical equivalent, 26mm or more of axial length.
* History of intraocular surgery.
* Presence of staphyloma.
* Other ocular diseases that could influence macular microstructure or visual function

Exit criteria:

* For reposition group, the patients will exit the research if the peeled ILM cannot reposition successfully.
* Due to adverse events, especially severe adverse events, the researchers consider withdrawal of patients based on concerns of safety and ethics;
* Drop out;
* The patients voluntarily withdraw the informed consent;
* Serious violation of the study protocol due to the subjects or investigators' reasons;
* Other reasons that the researchers believe for quitting the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity(BCVA) | Pre-operation and 6 months after operation
  Change from baseline BCVA at 6 months after operation, examined with snellen chart.

SECONDARY OUTCOMES:
Close rate of macular holes | 1 month after operation
  Observed from optical coherence tomography

OTHER OUTCOMES:
Morphologic changes of inner retina | 1，3，6 months after operation
  Dimpling observed from optical coherence tomography
Central retinal thickness change | Pre-operation and 1，3，6 months after operation
  Measured by software in optical coherence tomography
Mean foveal light sensitivity change | Pre-operation and 1，3，6 months after operation
  Measured by microperimetry
Fixation stability change | Pre-operation and 1，3，6 months after operation
  Measured by microperimetry
Multifocal electroretinogram(Mf-ERG) change | pre-operation and 1，3，6 months after operation
  An objective measurement of retinal functions
M-chart score change | Pre-operation and 1，3，6 months after operation
  M-horizontal score and M-vertical score
Visual function questionnaire-25(VFQ-25) score change | Pre-operation and 1，3，6 months after operation
  A questionnaire consisted of 25 visual function questions concerning life quality

CONTACTS AND LOCATIONS:
Overall Officials: Peiquan Zhao, PhD, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after the end of this clinical trails.The data included patients' serial number, gender, age, laterality and all outcome measurement
Supporting Information: Study Protocol, ICF
Time Frame: After enrollment completed; After the last followup of the last participant.

REFERENCES:
- [Derived] Tian T, Tan H, Zhu X, Zhang X, Zhao P. PEELED INTERNAL LIMITING MEMBRANE REPOSITION FOR IDIOPATHIC MACULAR HOLES: A Pilot Randomized Controlled Trial. Retina. 2023 Feb 1;43(2):191-199. doi: 10.1097/IAE.0000000000003645. Epub 2022 Oct 8. PMID 36695790